CLINICAL TRIAL: NCT05933720
Title: Evaluation of the Efficacy and Safety of the Drug Based on Vascular Regulatory Polypeptides for the Treatment of Patients With Lower Extremity Atherosclerotic Arterial Occlusive Disease.
Brief Title: Efficacy and Safety of the Regulatory Polypeptides in Patients With Peripheral Atherosclerosis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Principal Investigator, Lyasheva Anastasia Vladimirovna, Resident cardiovascular surgeon in the Department of Cardiovascular, Endovascular Surgery and Diagnostic Radiology, Ryazan State Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: Peripheral Arterial Disease; bypass grafting; polypeptides
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1; Peripheral Arterial Disease | interventions — Peptides

STUDY DESIGN:
Intervention Model Description: An open, prospective study is aimed at enrolling 120 patients with lower extremity atherosclerotic arterial occlusive disease. Patients are planned to undergo conservative therapy according to indications, including the use of a drug based on vascular polypeptides Slavinorm®, as well as a combination of conservative therapy, including a drug based on vascular polypeptides Slavinorm®, with surgical methods of treatment (femoral-popliteal bypass grafting with a synthetic graft above the knee). Subjects of similar age, gender, and ethnicity should be divided into four groups, respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients who undergo routine conservative treatment (Active Comparator): The patients who undergo routine conservative treatment for peripheral atherosclerotic occlusive disease as per clinical guidelines
  Interventions: Other: Routine conservative treatment
- Patients who undergo treatment with polypeptides (Experimental): The patients who undergo treatment with a complex of polypeptides isolated from the vessels of cattle is administered in / m, adults 1 vial (5 mg) 1 time / day 2 times a week. The course of treatment is 10 injections.
  Interventions: Drug: Polypeptides
- Patients who undergo femoral-popliteal bypass with a synthetic graft above the knee (Active Comparator): Patients who undergo the surgical method of treatment i.e. femoral-popliteal bypass grafting with a synthetic graft above the knee and routine conservative treatment as per clinical guidelines
  Interventions: Device: Femoral-popliteal bypass grafting with a synthetic graft above the knee; Other: Routine conservative treatment
- Patients who undergo femoral-popliteal bypass grafting and treatment with polypeptides (Experimental): Patients who undergo the surgical method of treatment i.e. femoral-popliteal bypass grafting with a synthetic graft above the knee with following treatment with a complex of polypeptides isolated from the vessels of cattle is administered in / m, adults 1 vial (5 mg) 1 time / day 2 times a week. The course of treatment is 10 injections.
  Interventions: Drug: Polypeptides; Device: Femoral-popliteal bypass grafting with a synthetic graft above the knee

INTERVENTIONS:
Drug: Polypeptides — The patients will undergo treatment with a drug based on vascular polypeptides Slavinorm®, a derivative from cattle vessels, registered in Russia for the treatment of patients with peripheral atherosclerotic occlusive disease.
  Other Names: vascular polypeptides Slavinorm®, a derivative from cattle vessels
  Arms: Patients who undergo femoral-popliteal bypass grafting and treatment with polypeptides; Patients who undergo treatment with polypeptides
Device: Femoral-popliteal bypass grafting with a synthetic graft above the knee — The patients with undergo an arterial revascularization - Femoral-popliteal bypass grafting with a synthetic graft above the knee
  Arms: Patients who undergo femoral-popliteal bypass grafting and treatment with polypeptides; Patients who undergo femoral-popliteal bypass with a synthetic graft above the knee
Other: Routine conservative treatment — The patients will undergo routine conservative treatment as per clinical guidelines (acetylsalicylic acid 100mg daily, atorvastatin 20mg daily)
  Arms: Patients who undergo femoral-popliteal bypass with a synthetic graft above the knee; Patients who undergo routine conservative treatment

SUMMARY:
The study is aimed at assessing the role of the activity of markers of endothelial dysfunction (cytotoxic malonic aldehyde (MDA), angiotensin II, endothelial nitric oxide synthase (NO), endothelin-1, prostacyclin) in the systemic circulation in patients with lower extremity atherosclerotic arterial occlusive disease undergoing open reconstructive interventions.

DETAILED DESCRIPTION:
The study will include 120 patients of similar age, gender, and ethnicity, they will be divided into four groups: Group I: 30 patients with lower extremity atherosclerotic arterial occlusive disease, stage IIA-IIB of the disease according to the Fontaine-Pokrovsky classification, receiving conservative therapy; Group II: 30 patients with lower extremity atherosclerotic arterial occlusive disease, stage IIA-IIB of the disease according to the Fontaine-Pokrovsky classification, receiving conservative therapy, including the drug based on vascular polypeptides Slavinorm®; Group III: 30 patients with lower extremity atherosclerotic arterial occlusive disease, stageIII-IV of the disease according to the Fontaine-Pokrovsky classification, receiving conservative therapy in combination with surgical methods of treatment (femoral-popliteal bypass grafting with a synthetic graft above the knee); Group IV: 30 patients with lower extremity atherosclerotic arterial occlusive disease, stage III-IV of the disease according to the Fontaine-Pokrovsky classification, receiving conservative therapy, including the drug based on vascular polypeptides Slavinorm®, in combination with surgical methods of treatment (femoral-popliteal bypass grafting with a synthetic graft above the knee).

ELIGIBILITY:
Inclusion Criteria:

men or women over 18 years of age with lower extremity atherosclerotic arterial occlusive disease, confirmed with instrumental work-up methods (ultrasonography or angiography).

Exclusion Criteria:

men or women under 18 years of age; history of anaphylaxis; hypersensitivity to any of the components that make up the drug Slavinorm®, and proteins of animal origin; absolute and relative contraindications to the treadmill test; failure to walk at a minimum speed of 3.2 km/h (2 mph) at a minimum treadmill angle for at least 2 minutes during the stress test during the screening phase; depression of the ST segment more than 1 mm in one or more standard leads on the electrocardiogram; peripheral artery disease not associated with atherosclerosis; patients who underwent reconstructive surgery or invasive interventions on the arteries of the lower extremities in history without a clinic of intermittent claudication; angina pectoris III-IV functional class (FC) according to the CCS classification; body mass index >35 kg/m2; acute or chronic renal (creatinine clearance less than 30 ml / min) and / or liver failure [aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 3 times the upper limit of normal]; chronic heart failure III-IV FC according to NYHA; acute coronary syndrome within 6 months. before the start of the screening period; any clinically significant condition or comorbidity that, in the opinion of the Investigator, would preclude the patient from participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Lower artery or bypass graft thrombosis | 1 year
  The rate of the Lower artery or bypass graft thrombosis
disease progression | 1 year
  The rate of the disease progression
restenosis | 1 year
  Restenosis rate

SECONDARY OUTCOMES:
limb loss | 1 year
  Limb loss rate
changes in pain-free walking distance | 1 year
  Changes in the parameter of pain-free walking distance (in meters)
changes in ankle-brachial index | 1 year
  Changes in the parameter of ankle-brachial index measured at rest

CONTACTS AND LOCATIONS:
Overall Officials: Igor Suchkov, Study Chair — Ryazan State Medical University
Locations (1):
- RyazanSMU, Ryazan, Russia